CLINICAL TRIAL: NCT05399992
Title: VICTORION REAL: An International Prospective Real-world Study to Evaluate the LDL-C changE and Adherence to incLisiran in Participants With Primary Hypercholesterolemia or Mixed Dyslipidemia
Brief Title: Study Evaluating LDL-C Change and Adherence to Inclisiran Lipid-lowering Therapy in ASCVD
Acronym: VICTORION REAL
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839A12401
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
Keywords: primary hypercholesterolemia; mixed dyslipidemia; real-world study; inclisiran; lipid-lowering therapy; LLT; ASCVD
MeSH Terms: interventions — ALN-PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Inclisiran cohort: Participants prescribed inclisiran alone or with other LLTs as per approved label
  Interventions: Other: Inclisiran

INTERVENTIONS:
Other: Inclisiran — Prospective observational study. There is no treatment allocation. Patients who are eligible to receive inclisiran will be enrolled into this study.

SUMMARY:
This observational prospective study aims to evaluate the LDL-C change and adherence to inclisiran in combination with other lipid lowering therapies or lipid lowering treatments (LLTs) under conditions of routine clinical practice.

DETAILED DESCRIPTION:
Patients will be enrolled over a period of 23 months, and followed for up to 24 months to assess for study outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are 18 years or older
2. Participants with hypercholesterolemia having a diagnosis of ASCVD, ASCVD RE or HeFH
3. Participants who are not at LDL-C goal as per their CV risk according to respective clinical guidelines
4. Participants who per physician's criteria need to optimize their LLT
5. Participants who provide written informed consent to participate in the study
6. Participants who initiate inclisiran under conditions per local label and have LDL-C values available at baseline or within 3 months before treatment initiation.

Exclusion Criteria:

1. Participants that have received inclisiran previously
2. Participants participating in a clinical trial with investigational product 3 Participants switching from previous PCSK9 mab treatment (within 90 days prior to Index date)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult participants with an underlying diagnosis of Atherosclerotic Cardiovascular Disease (ASCVD), ASCVD risk equivalent (ASCVD RE), or Heterozygous familial hypercholesterolemia (HeFH) and elevated levels of Low density lipoprotein - Cholesterol (LDL-C)
Sampling Method: Non-Probability Sample
Enrollment: 847 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Percentage change in LDL-C from baseline to 10 months | Baseline, 10 months
  Percentage change in Low density lipoprotein - Cholesterol (LDL-C)

SECONDARY OUTCOMES:
Percentage change in LDL-C from baseline | Baseline, month 4, month 16, month 22
  Percentage change in LDL-C from baseline is collected
Percentage change in LDL-C from baseline by ≥50% | Month 4, month 10, month 16, month 22
  Percentage change in LDL-C from baseline by ≥50%
Percentage change in LDL-C from baseline by ≥30% | Month 4, month 10, month 16, month 22
  Percentage change in LDL-C from baseline by ≥30%
Proportion of participants achieving LDL-C<55 mg/dL | Proportion of participants achieving LDL-C<55 mg/dL Month 4, month 10, month 16 and month 22
  Proportion of participants achieving LDL-C<55 mg/dL
Proportion of participants achieving LDL-C<70 mg/dL | Month 4, month 10, month 16 and month 22
  Proportion of participants achieving LDL-C<70 mg/dL
Time-averaged percentage change in LDL-C from baseline | Baseline, month 4, month 10, month 16 and month 22
  Time-averaged percentage change in LDL-C from baseline
Proportion of participants achieving ≥50% reduction in LDL- C at month 10 and maintaining this at 16, 22 and 24 months | Month 10, month 16, month 22 and month 24
  Proportion of participants achieving ≥50% reduction in LDL C at month 10 and maintaining this at 16, 22 and 24 months
Proportion of participants achieving ≥30% reduction in LDL C from baseline to 10 months and maintaining until 24 months | Baseline, month 10, month 24
  Proportion of participants achieving ≥30% reduction in LDL C from baseline to 10 months and maintaining until 24 months
Proportion of participants achieving <55 mg/dL and <70 mg/dL in LDL-C at 10 months and maintaining until 24 months | Month 10 and month 24
  Proportion of participants achieving <55 mg/dL and <70 mg/dL in LDL-C at 10 months and maintaining until 24 months
Inclisiran cohort : Percentage of days covered by inclisiran | 12 months and 24 months
  Inclisiran cohort : Percentage of days covered by inclisiran
Inclisiran cohort : Mean PDC | 12 months and 24 months
  Mean Proportion of Days Covered (PDC) for inclisiran cohort is collected
Inclisiran cohort : Proportion of participants with a PDC ≥ 80% | 12 months and 24 months
  Proportion of participants with a PDC ≥ 80% (sensitivity: 90%/100%)
Proportion of participants remaining on initial baseline therapy | Baseline, month 12 and month 24
  Proportion of patients remaining on initial baseline therapy in the inclisiran cohort
Time to discontinuation of any newly initiated therapies | Month 12 and month 24
  Time to discontinuation of any newly initiated therapies
Time to discontinuation of any newly initiated therapies by specific LLT | Month 12 and month 24
  Time to discontinuation of any newly initiated therapies by specific LLT
Change from baseline in scores from the TSQM (modified) instrument | Baseline, month 12 and month 24
  The 14-item Treatment Satisfaction Questionnaire for Medication (TSQM) version 1.4 is an instrument to assess patients' satisfaction with medication, providing scores on four scales - side effects, effectiveness, convenience and global satisfaction.
  TSQM V1.4 has a score range of 0 to 100 with with higher scores indicating higher patient satisfaction with medication.
Descriptive adherence data based on Adherence AAQ | Month 12 and month 24
  Adherence Assessment Questionnaires (AAQ) measures the degree of identified non-adherence to LLT therapy.
  AAQ has a score range from 0 (not adherent at all) to 100 (absolute adherent).
Descriptive adherence data based on ABQ | Month 12 and month 24
  Adherence Barriers Questionnaire (ABQ) is an instrument for identifying specific barriers to medication-related adherence.
  ABQ is a descriptive analysis. The number and proportion of patients affected by each barrier will be reported for inclisiran participants.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- Austria (5):
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Sankt Veit im Pongau
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Shenzhen, Guangdong, China
- Israel (3):
  - Novartis Investigative Site, Holon, Gush Dan
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Malaysia (2):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kuala Lumpur
- Saudi Arabia (3):
  - Novartis Investigative Site, Riyadh, Saudi
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Tabuk
- Switzerland (7):
  - Novartis Investigative Site, Fribourg, CH
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Olten
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- United Arab Emirates (5):
  - Novartis Investigative Site, Abu Dhabi, Abu Dhabi Emirate
  - Novartis Investigative Site, Dubai, United Arab Emirates
  - Novartis Investigative Site, Abu Dhabi
  - Novartis Investigative Site, Al Ain City
  - Novartis Investigative Site, Dubai
- United Kingdom (12):
  - Novartis Investigative Site, High Wycombe, Buckinghamshire
  - Novartis Investigative Site, Louth, Lincolnshire
  - Novartis Investigative Site, Sunderland, Tyne and Wear
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Bromwich
  - Novartis Investigative Site, Burton-on-Trent
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, Lancaster
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Middlesex